CLINICAL TRIAL: NCT05920538
Title: Effects of Subcutaneously Infiltrated Nicardipine on the Success Rate of Radial Artety Cannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 764/2565(IRB3)
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Radial Artery Cannulation
Keywords: Nicardipine; radial artery; artery cannulation; ultrasound
MeSH Terms: interventions — Nicardipine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicardipine (Experimental): Using nicardipine 0.5 mg(0.5ml) subcutaneously infiltrated by ultrasound before redial artery cannulation.
  Interventions: Drug: Nicardipine
- Normal saline (Placebo Comparator): Using normal saline 0.5ml subcutaneously infiltrated by ultrasound before redial artery cannulation
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Nicardipine — Subcutaneous infiltrate drug at puncture site by ultrasound-guided
  Arms: Nicardipine
Other: Normal saline — Subcutaneous infiltrate NSS at puncture site by ultrasound-guided
  Arms: Normal saline

SUMMARY:
The goal of this study is to compare the success rate of subcutaneously infiltrated nicardipine to normal saline in radial artery cannulation

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* the patient who need to arterial line

Exclusion Criteria:

* allergy to nicardipine
* history of peripheral artery disease
* BMI > 40 kg/m2
* unwilling to participate or denial of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of radial artery cannulation since first skin puncture | 10 minute from puncture at skin
  Success rate of radial artery cannulation since first skin puncture

SECONDARY OUTCOMES:
radial artery diameter | Pre-induction to 3 minute after subcutaneous infiltration
  Pre-induction radial artery diameter, post-induction radial artery diameter, radial artery diameter after subcutaneous infiltration at 0,1,2 and 3 minute
Time from first skin puncture to success cannulation | 10 minutes
  Time from first skin puncture to present of arterial wave form, assessed less than 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Phuriphon Songarj, MD, Study Director — Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand
Locations (1):
- Anesthesiology Department, Bangkok, Thailand